CLINICAL TRIAL: NCT02471209
Title: Biliary Atresia, Hepatic Buffer Response and Sevoflurane
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: mzk-0003-2011
Record Dates: First submitted 2015-06-03; First posted 2015-06-15 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Biliary Atresia
MeSH Terms: conditions — Biliary Atresia | interventions — Sevoflurane; Anesthesia, General

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biliary Atresia Infants: Twenty-five infants diagnosed with Biliary Atresia and undergoing surgery were included in the study (age range 1-3 months). Inclusion criteria were persistent yellow skin or sclera, pale stool (in severe cases, clay-like), and hepatomegaly; increased serum bilirubin (progressively or no decline after increase), increased total bilirubin (TBil) dominated by increased direct bilirubin (DBil) (>60%); elevated liver enzymes; ultrasound confirmation of poor gallbladder filling and signs of liver fibrosis; with radionuclide imaging confirmation of obstructed biliary excretion. Infants were excluded if they had concomitant cardiovascular or abdominal organ malformations.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Sevoflurane — general anesthesia with 2% followed by 3% sevoflurane
  Other Names: general anesthesia

SUMMARY:
To evaluate the effects of sevoflurane on hepatic blood flow (HBF) and hepatic arterial buffer response (HABR) in infants with obstructive jaundice by Doppler ultrasound.Twenty-five infants with biliary atresia (1-3 months-of-age) scheduled for a Kasai procedure were enrolled. portal vein blood flow (PBF), hepatic arterial blood flow (HABF) and hepatic blood flow (HBF) were measured by Doppler ultrasound before induction, and after inhalation of 2 and 3% sevoflurane.

DETAILED DESCRIPTION:
Children suffering from hepatobiliary disease also have an hepatic arterial buffer response (HABR) with reduced portal vein blood flow (PBF) and compensatory increases in hepatic arterial blood flow (HABF) which can help maintain hepatic blood flow (HBF). For infants with obstructive hepatobiliary disease, reduced HBF may affect drug metabolism and increase the risk of respiratory depression during analgesia, which can be life-threatening.

To evaluate the effects of sevoflurane on HBF and HABR in infants with obstructive jaundice by Doppler ultrasound.Twenty-five infants with biliary atresia (1-3 months-of-age) scheduled for a Kasai procedure were enrolled. PBF, HABF and HBF were measured by Doppler ultrasound before induction, and after inhalation of 2 and 3% sevoflurane.

ELIGIBILITY:
Inclusion Criteria:

* persistent yellow skin or sclera, pale stool (in severe cases, clay-like), and hepatomegaly;
* increased serum bilirubin (progressively or no decline after increase), increased total bilirubin (TBil) dominated by increased direct bilirubin (DBil) (>60%);
* elevated liver enzymes;
* ultrasound confirmation of poor gallbladder filling and signs of liver fibrosis;
* with radionuclide imaging confirmation of obstructed biliary excretion

Exclusion Criteria:

* concomitant cardiovascular or abdominal organ malformations

Ages: 1 Month to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infants with biliary atresia scheduled for a Kasai procedure
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2012-01; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
portal blood flow | 10 minutes
hepatic arterial blood flow | 10 minutes
hepatic blood flow | 10 minutes

SECONDARY OUTCOMES:
blood pressure | 5 minutes
  noninvasive blood pressure
renal blood flow | 10 minutes
femoral vein blood flow | 10 minutes